CLINICAL TRIAL: NCT04652765
Title: COMBO Trial: Camostat With Bicalutamide for COVID-19
Brief Title: Camostat With Bicalutamide for COVID-19
Acronym: COMBO
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI Decision to close/stop the study due to no new accrual.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COV2005; IRB00254142 (Other: JHM IRB)
Record Dates: First submitted 2020-12-02; First posted 2020-12-03 (Actual); Results first posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Covid19; SARS-CoV Infection; Coronavirus Infection
Keywords: COVID-19; Coronavirus; Camostat; bicalutamide; TMPRSS2; SARS-COV-2
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections | interventions — camostat; bicalutamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Standard of care (SOC) (No Intervention): SARS-CoV-2 positive participants will receive SOC therapy alone.
- SOC plus camostat (Active Comparator): SARS-CoV-2 positive participants will receive SOC therapy as well as camostat for 7 days.
  Interventions: Drug: Camostat Mesilate
- SOC plus camostat and bicalutamide (Active Comparator): SARS-CoV-2 positive participants will receive SOC therapy as well as camostat and bicalutamide for 7 days.
  Interventions: Drug: Camostat Mesilate; Drug: Bicalutamide 150 mg

INTERVENTIONS:
Drug: Camostat Mesilate — Camostat 600mg by mouth four times a day, for a total of 7 days
  Other Names: camostat
  Arms: SOC plus camostat; SOC plus camostat and bicalutamide
Drug: Bicalutamide 150 mg — Bicalutamide 150mg by mouth once daily, for a total of 7 days
  Arms: SOC plus camostat and bicalutamide

SUMMARY:
This will be a randomized, open-label study to determine if camostat+ bicalutamide decreases the proportion of people with COVID-19 who require hospitalization, compared to historical controls. Patients with symptomatic COVID-19, diagnosed as outpatients, will be randomized 1:1, stratified by gender, to treatment with standard of care alone (Arm 1) or with camostat and bicalutamide (Arm 2).

ELIGIBILITY:
Inclusion Criteria:

* >= 60 years of age
* COVID-19 infection, confirmed by polymerase chain reaction (PCR) test <=5 days from enrollment done in the ambulatory setting
* Able to provide informed consent
* Symptom related to COVID-19. This includes: fever or chills, cough, shortness of breath or difficulty breathing, fatigue, muscle or body aches, headache, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting, diarrhea or other symptom recognized by the Centers for Disease Control to be a symptom of COVID-19.

Exclusion Criteria:

* Patients who undergo asymptomatic screening test that is positive and remain asymptomatic during the eligible time window
* Patients who have had one or more positive more than 5 days prior to enrollment but within 60 days of enrollment (ex. if a patient has a positive test 10 days prior to enrollment and then a second positive test the day referred for enrollment, that patient would be excluded. If a patient had a positive test 5 months ago, and then another positive test the day he/she was referred for enrollment, that patient would be eligible)
* Unable to take oral medication
* Male patients with female partners of reproductive potential who are unable to maintain effective contraception during the recommended time period (during treatment and for 130 days after the final dose)
* Symptoms requiring hospitalization or immediate referral to hospital
* Taking bicalutamide, any systemic hormonal therapy, or camostat within one month of study entry
* Known hypersensitivity to bicalutamide, or camostat, or its components.
* On coumadin anticoagulation (because of drug-drug interaction with bicalutamide)
* Self-reported past medical history of chronic liver disease or cirrhosis
* Self-reported myocardial infarction within 6 months or past medical history of congestive heart failure with known ejection fraction < 40%
* Taking any other investigational treatment for COVID-19 or COVID-19 prophylaxis (COVID-19 vaccines and treatments allowed under FDA Emergency Use Authorization are allowed.)

Women and people from all ethnic and race groups are eligible for this study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine H Marshall, MD/MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Started | 1 | 2 | 3
Completed | 1 | 2 | 2
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide | Total
Number analyzed (Participants) | 1 | 2 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3 | 6
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 61 [61 to 61] | 62.5 [60 to 65] | 61 [60 to 62] | 61.5 [60 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 2 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 2 | 3
  White | 1 | 1 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Hospitalization
Description: Number of outpatient participants diagnosed with COVID-19 who require hospitalization by day 28
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Number analyzed (Participants) | 1 | 2 | 3
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants Experiencing Symptoms
Time Frame: up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Number analyzed (Participants) | 1 | 2 | 2
Participants | 1 | 2 | 2

3. Secondary Outcome: Number of Drug-related Adverse Events
Description: Number of adverse events, as defined by NCI CTCAE version 5.0, that are related to the study drug (or therapy)
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Number analyzed (Participants) | 1 | 2 | 2
Participants | 0 | 0 | 1

4. Secondary Outcome: Number of Drug-related Serious Adverse Events
Description: Number of serious adverse events, as defined by NCI CTCAE version 5.0, that are related to the study drug (or therapy)
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Number analyzed (Participants) | 1 | 2 | 2
Participants | 0 | 0 | 0

5. Secondary Outcome: All-cause Mortality
Description: Number of participants deceased.
Time Frame: up to 60 days
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
Number analyzed (Participants) | 1 | 2 | 2
Participants | 0 | 0 | 0

6. Other Pre Specified Outcome: Duration of Hospitalization
Description: Number of calendar days in the hospital
Time Frame: up to 60 days
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Participants Requiring Upgrade to Intermediate Care Unit (IMC)
Time Frame: up to 60 days
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Duration of IMC Stay
Description: Number of calendar days in IMC unit
Time Frame: up to 60 days
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Number of Participants Requiring Upgrade to Intensive Care Unit (ICU)
Time Frame: up to 60 days
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Duration of ICU Stay
Description: Number of calendar days in ICU
Time Frame: up to 60 days
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Number of Participants Requiring Mechanical Ventilation
Time Frame: up to 60 days
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Duration on Mechanical Ventilation
Description: Number of calendar days requiring mechanical ventilation
Time Frame: up to 60 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 60 days
Description: Only non COVID-19 adverse event were collected
Arm/Group | Standard of Care (SOC) | SOC Plus Camostat | SOC Plus Camostat and Bicalutamide
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care (SOC) (N=1) | SOC Plus Camostat (N=2) | SOC Plus Camostat and Bicalutamide (N=3)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04652765/Prot_SAP_000.pdf